CLINICAL TRIAL: NCT03480620
Title: Access to an Online Telerehabilitation Exercise Program Post-discharge From a Comprehensive Pain Management Program: Patient Acceptance and Impact on Outcomes Sustainability and Return to Opioid Use
Brief Title: Post Discharge Online Telerehabilitation Program
Acronym: OTP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Brooks Rehabilitation (Other)
Collaborators: Florida Physical Therapy Association (Unknown); Yoga, Fitness, Mindfulness (Unknown); ReadyOp (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BRCRC2017_001
Record Dates: First submitted 2018-02-02; First posted 2018-03-29 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pain, Chronic
Keywords: Telehealth; Telerehabilitation; Chronic pain; Post-discharge care
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: A stratified random sampling approach will be used for this study whereby graduates from the BPRP will first be identified as having weaned off opioid medications (weaners) or did not wean off opioid medication (non-weaners). Once stratified into these two groups, participants will then be randomly assigned to either the standard care group (control group) or the telerehabilitation group (intervention group) based on sequential enrollment into each study group. Participants will continue with there post-discharge exercise and self-management program for one year, completing follow up assessment using the online platform at 1, 3, 6, 9, and 12 months post discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Participant randomized into the telerehabilitation group will receive verbal and written discharge recommendations from each member of the team as usual. They will also be given a login to the online telerehabilitation platform where they will find the designated flexibility routines which can be accessed from a computer, tablet/slate, or smart phone at any time. Participant will receive electronic reminders via email and/or text message to perform their home program and complete the follow up questionnaires. Other physical therapy exercises may be recommended based on individual patient's need. These exercises will be provided in verbal and written form.
  Interventions: Other: Online Telerehabilitation Platform Access
- Usual care (Active Comparator): Participants randomized into the usual care group will receive verbal and written discharge recommendations from each member of the team as usual. They will be provided with a copy of the DVD and instructed to practice one of the two routines at least 5 days per week. They will also be given a login to the online platform but will only have access to complete the follow up questionnaires. Participant will receive electronic reminders via email and/or text message to complete the follow up questionnaires. Other physical therapy exercises may be recommended based on individual patient's need. These exercises will be provided in verbal and written form.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Online Telerehabilitation Platform Access — Participants will have 24/7 access to a standardized set post-discharge exercise videos and self-management instructions across multiple internet connected devices (e.g. computer, tablet, smartphone). Standardized exercises include a flexibility routine that participants learned and performed with a physical therapist while in the pain management program. Self-management instructions are also written versions of concepts learned and practiced with a member of the multidisciplinary team during the pain management program.
  Arms: Telerehabilitation
Other: Usual care — Participants are given a DVD of the standardized post-discharge exercise videos and a written copy of the self-management instructions as described in the experimental group.
  Arms: Usual care

SUMMARY:
This study will evaluate the sustainability of pain and functional outcomes along with return to opioid use in a population of patients that successfully completed a comprehensive interdisciplinary pain rehabilitation program. In addition, this study will compare outcomes sustainability and return to opioid use between pain program graduates who receive post discharge self-management resources consisting of a DVD with videos of recommended flexibility practice (standard of care) or access to an online telerehabilitation platform that provides patients with access to the flexibility practice videos on a variety of telecommunication devices (e.g., computer, smart phone, tablet).

DETAILED DESCRIPTION:
The primary purpose of this paper is to compare the use of an online telerehabilitation platform versus a standard prerecorded DVD in supporting the sustainability of outcomes achieved during a comprehensive multidisciplinary pain rehabilitation program.

Primary Hypotheses Graduates from a comprehensive interdisciplinary pain rehabilitation program will…

1. …demonstrate greater adherence to post-discharge home exercise recommendations when given access to an online telerehabilitation platform compared to DVDs offered as current standard of care.
2. …achieve greater sustainability of programs outcomes including pain intensity, level of function, and reduction of opioid use.

Primary Research Questions

1. Does access to an online telerehabilitation platform impact adherence to post-discharge home exercise recommendations in graduates from a comprehensive interdisciplinary pain rehabilitation program?
2. Does access to an online telerehabilitation platform impact outcomes sustainability and opioid use in graduates from a comprehensive interdisciplinary pain management program?

Additional items that will be evaluated by this study include the participants' experience and satisfaction with use of the online telerehabilitation platform.

Secondary Hypotheses

1. Participants using the online telerehabilitation platform will report a more enjoyable experience and overall greater satisfaction with post-discharge self-management compared to participants receiving standard of care.
2. Utilization of the online telerehabilitation platform will be associated with perceptions of usefulness and ease of use of internet technology.

Secondary Research Questions

1. Does use of an online telerehabilitation platform impact patient satisfaction with post-discharge self-management compared to current standard of care?
2. Does internet technology acceptance impact utilization of post-discharge self-management resources provided through an online telerehabilitation platform?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pain consistent with IASP definition.
* Classification as a "completer" of the Brooks Rehabilitation Pain Rehabilitation Program by attending the expected number of sessions and achieving at least 90% of goals.
* Able to read, write, and understand spoken English fluently.

Exclusion Criteria:

* Any medical condition that would place the participant at risk with performing a home exercise program.
* Inability to see or hear the audio visual device from a distance of at least 5 feet (may use headphones).
* Cognitive impairment or learning barriers preventing appropriate ability to access and navigate the study-related web-site or play the study-related DVD's.
* Lack of regular access to internet service.
* Lack of regular access to an internet connected audio-visual device (e.g., smartphone, computer, tablet, etc) in a location with sufficient space to perform exercises.
* Not familiar with basic internet navigation (i.e. able to locate and access a desired website and use basic within-site navigation tools such as scrolling and clicking on links.
* Currently pregnant (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence to post-discharge home exercise recommendations | 12 months post discharge
  Self-reported home exercise program adherence. Utilization data from the online telerehabilitation platform will also be collected for the telerehabilitation group.
PROMIS Measure - Physical Function - Short Form 8b | 12 months post discharge
  PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living, such as running errands. A single Physical Function capability score is obtained from a short form. Each Physical Function instrument is appropriate for the adult general population and adults with chronic health conditions.
PROMIS Measure - Pain Interference - Short Form 4a | 12 months post discharge
  The PROMIS Pain Interference item banks assess self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Pain Interference also incorporates items probing sleep and enjoyment in life, though the item bank only contains one sleep item. The pain interference short forms are universal rather than disease-specific. All assess pain interference over the past seven days.
PROMIS Measure - Self-Efficacy for Managing Symptoms - Short Form 8a | 12 months post discharge
  Self-efficacy is defined as confidence in one's ability to successfully perform specific tasks or behaviors. Self-Efficacy for Managing Chronic Conditions assesses confidence in one's ability to successfully perform specific tasks or behaviors related to one's health in a variety of situations. Several domains of Self-Efficacy for Managing Chronic Conditions relate to specific aspects of managing chronic conditions.
  Self-Efficacy for Managing Chronic Conditions - Manage Symptoms: Confidence to manage/control their symptoms, to manage their symptoms in different settings and to keep symptoms from interfering with work, sleep, relationships or recreational activities.
  The Self-Efficacy item banks are universal rather than disease-specific. The respondent should be an adult (age18+) and have at least one chronic health condition. The PROMIS Adult Self-Efficacy items banks have been modified from the NIH Toolbox Self-Efficacy item bank.
PROMIS Measure - Self-Efficacy for Managing Emotions - Short Form 8a | 12 months post discharge
  Self-efficacy is defined as confidence in one's ability to successfully perform specific tasks or behaviors. Self-Efficacy for Managing Chronic Conditions assesses confidence in one's ability to successfully perform specific tasks or behaviors related to one's health in a variety of situations. Several domains of Self-Efficacy for Managing Chronic Conditions relate to specific aspects of managing chronic conditions.
  Self-Efficacy for Managing Chronic Conditions - Manage Emotions: Confidence to manage/control symptoms of anxiety, depression, helplessness, discouragement, frustration, disappointment and anger.
  The Self-Efficacy item banks are universal rather than disease-specific. The respondent should be an adult (age18+) and have at least one chronic health condition. The PROMIS Adult Self-Efficacy items banks have been modified from the NIH Toolbox Self-Efficacy item bank.

SECONDARY OUTCOMES:
Technology Acceptance Model Questionnaire | 12 months post discharge
  The Technology Acceptance Model (TAM) Questionnaire used in this study is a 23-item self report questionnaire investigating participants perceived usefulness (PU) and perceived-ease-of-use (PEOU) of the internet. Higher scores for PU and PEOU are purported to influence an individual's intention to use a particular technology.
Patient Satisfaction | 12 months post discharge
  A single item rating satisfaction with home exercise and self-management program

OTHER OUTCOMES:
Program-Specific Outcomes Questionnaire | 12 months post discharge
  A 33-item questionnaire developed by the pain program to track post-discharge outcomes over time. This measure will be compared to the PROMIS measures to evaluate concurrent validity of the program-specific questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooks Rehabilitation, Jacksonville, Florida, United States